CLINICAL TRIAL: NCT02336867
Title: Therapeutic Management of Complex Anal Fistulas by Installing a Closure Clip: Multicentre Randomized Controlled Trial
Acronym: FISCLOSE
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHU-2018; 2014-A00441-46 (Registry Identifier: 2014-A00441-46)
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Complex Anal Fistula
Keywords: Complex anal fistula, clip,

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Experimental group (Experimental): closure clip (OTSC® Proctology Laboratory: OVESCO and French Distributor: Life Partners)
  Interventions: Device: Closure clip (OTSC® Proctology)
- Control group (Other): advancement flap technique
  Interventions: Device: Closure clip (OTSC® Proctology)

INTERVENTIONS:
Device: Closure clip (OTSC® Proctology)

SUMMARY:
Anal fistulas are the main etiology of perianal abscesses and suppurations. They are common and generally associated with pain, anal incontinence, impaired quality of life and work incapacity. The therapeutic management of this disease has a double objective: heal the suppuration and preserve the sphincter function. Each year, anal fistulas affect 1 in 10 000 in the normal population, with a difference in prevalence between men and women (1.23 per 10 000 men and 0.56 per 10 000 women). The average age of the patients was 40 years (Simpson et al., 2012).

In about 80% of cases, anal fistulas are secondary to an infection of Hermann and Desfosses' anal glands (cryptogenic or cryptoglandular). Infection of the anal gland can result in an abscess between the internal and external sphincters, which in turn can spread to other parts of the perianal region. The infection can follow many directions from this point in the intersphincteric plan. When the pus reaches the skin, the fistula is formed. Anal fistula therefore has always an intraductal origin, cryptic, with a primary port at this level, and the disregard of which causes the recurrence of the fistula; and usually a secondary port in the skin.

Fistulas are usually divided into two groups. The first group contains fistulas called "simple", which are intersphincteric fistulas or trans-sphincteric involving only the lower third of the sphincter complex. Fistulas usually didn't affect any muscle. The second group contains fistulas called "complex". These are intersphincteric, trans-sphincteric, or even suprasphincteric, extrasphincteric fistulas.

For many years, the treatment of choice was to open the fistula (fistulotomy), but this procedure was associated with a risk of incontinence, the consequences could be potentially devastating. Other surgical treatments include setons, fibrin glue, collagen plugs and advancement flap technique to cover internal opening of the fistula. The success of these therapies remains variable.

The advancement flap technique remains a strategy of choice in the treatment of anal fistulas and particularly in the case of complex fistulas. The success rate of the advancement flap technique remains variable across studies but a recent meta-analysis finds a success rate of around 60%.

A new technique for closing anal fistula is currently in development with the use of a closure clip nitinol (OTSC® Proctology Laboratory: OVESCO and French Distributor: Life Partners). This new technique has been validated in a porcine model of anal fistula, ensuring the safety of the device. A first case was published in a patient with complex anal fistula (high trans-sphincteric). After erosion fistula tract with a special brush, a nitinol clip (OTSC® Proctology) was deposited on the internal opening of the fistula. Eight months after surgery, the fistula was healed and the clip was removed by cutting with special pliers. This technique is currently being broadcast and dozens of patients were treated with this clip without any further scientific validation of the process.

To date, this innovative technique of the closure clip has not yet been assessed in a randomized controlled trial. It is therefore essential to carry out a prospective evaluation in order to determine the effectiveness and safety of this new device in the case of complex anal fistulas.

DETAILED DESCRIPTION:
After validation of the inclusion and exclusion criteria, the patients included in this clinical trial will be randomized between the two arms of the study for the closure of the anal fistula:

* Control group: advancement flap technique Experimental group: closure clip (OTSC® Proctology Laboratory: OVESCO and French Distributor: Life Partners)

Follow up of the patients will be performed until 1 year after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Complex anal fistula (intersphincteric, trans-sphincteric, or even suprasphincteric, extrasphincteric) drained and requiring closing intervention of fistula.
* Obtaining the patient's written consent
* Naive patient to any surgical treatment for fistula closure
* Patient receiving a social security scheme

Exclusion Criteria:

* <18 years and> 80 years
* BMI> 35 kg / m²
* Rectovaginal or rectourethral fistulas
* Infections : sepsis, tuberculosis or HIV
* History of allergy to nickel
* Cognitive disorders or major disability making it impossible to understand the study and signed an informed consent
* Already included in another clinical trial patients
* breastfeeding or pregnancy
* Legal incapacity (person deprived of liberty or guardianship)
* Patients not compliant with the criteria of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with healed anal fistula | at 3 months after surgery
  The diagnosis will be made by the lack of leakage alleged by the patient for at least one month and found on clinical examination

SECONDARY OUTCOMES:
Anal fistula healing | at 6 months and 1 year
VAS proctologic pain | days 0, 1, 2, 3, 15, 30, 60, 90, 180 and 365
Anal incontinence score (questionnaire Jorge and Wexner) | days 0, 15, 30, 60, 90, 180 and 365
Digestive disorders and quality of life (GIQLI questionnaire) | days 0, 15, 30, 60, 90, 180 and 365
Quality of life (EQ5D Questionnaire) | days 0, 30, 90, 365

CONTACTS AND LOCATIONS:
Overall Officials: Anne DUBOIS, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Dubois A, Carrier G, Pereira B, Gillet B, Faucheron JL, Pezet D, Balayssac D. Therapeutic management of complex anal fistulas by installing a nitinol closure clip: study protocol of a multicentric randomised controlled trial--FISCLOSE. BMJ Open. 2015 Dec 16;5(12):e009884. doi: 10.1136/bmjopen-2015-009884. PMID 26674505